CLINICAL TRIAL: NCT04211090
Title: A Phase II Study to Evaluate Camrelizumab With Pemetrexed / Carboplatin in Patients With Brain Metastases of Driven Gene-negative, Non-squamous Non-small Cell Lung Cancer
Brief Title: Camrelizumab With AC in Patients With Brain Metastases of Driven Gene-negative,NSCLC
Acronym: CAP-BRAIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li-kun Chen, director physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-203-X04
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Non-squamous Non-small-cell Lung Cancer; Brain Metastases
Keywords: Non-squamous Non-small-cell Lung Cancer; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — camrelizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Intervention Model Description: patients with brain metastases of driven gene-negative, non-squamous non-small cell lung cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab with pemetrexed / carboplatin (Experimental): Camrelizumab with pemetrexed / carboplatin in patients with brain metastases of driven gene-negative, non-squamous non-small cell lung cancer
  Interventions: Drug: Camrelizumab; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab with pemetrexed / carboplatin in patients with brain metastases of driven gene-negative, non-squamous non-small cell lung cancer, Participants receive a 3-week cycle (Q3W) treatment，Treatment continued until disease progression or unacceptable toxicity or death or, for the immunotherapy regimens
Drug: Pemetrexed — Camrelizumab with pemetrexed / carboplatin in patients with brain metastases of driven gene-negative, non-squamous non-small cell lung cancer, Participants receive a 3-week cycle (Q3W) treatment，Treatment continued until disease progression or unacceptable toxicity or death or, for the immunotherapy regimens
Drug: Carboplatin — Camrelizumab with pemetrexed / carboplatin in patients with brain metastases of driven gene-negative, non-squamous non-small cell lung cancer, Participants receive a 3-week cycle (Q3W) treatment，Treatment continued until disease progression or unacceptable toxicity or death or, for the immunotherapy regimens

SUMMARY:
The primary hypothesis is that camrelizumab in combination with pemetrexed/ carboplatin will present a better efficacy for treatment of first line metastatic non-squamous non-small cell lung cancer and minimize the risk of toxicity

DETAILED DESCRIPTION:
This is a prospective, open-label, phase Ⅱ studyto evaluate the efficacy and safetyof camrelizumab combined with pemetrexed/ carboplatin in participants with brain metastases ofnon-squamous non-small cell lung cancer.Paticipant was confirmed without EGFR activating mutation or ALK fusion, and received no prior systemic therapy.Patients would receive camrelizumab in combination with pemetrexed/ carboplatin for 4 cycles，followed by camrelizumab and pemetrexed as maitenance treatment until progression, camrelizumab will be administered no more than 24 months. PD-L1 expression assessed with 22C3 pharmDx assay will be used as a stratification factor.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of non-squamous non-small cell lung cancer（NSCLC）
2. Patients with asymptomatic BM or intracranial hypertension symptoms can be controlled after dehydration therapy, who can continue medication to maintain stable symptoms at enrollment or during the study;
3. Patients with MRI confirmed parenchymal brain metastases with ≥ 3 brain lesions; or patients with 1-2 brain lesions who are not suitable for or refuse local therapy. At least one measurable lesion must be ≥ 5 mm in diameter in brain lesions; patients with local meningeal metastases are allowed to be included, but those with extensive meningeal metastases are not included;
4. No prior systemic therapy for metastatic NSCLC; chemotherapy and/or radiotherapy as part of neoadjuvant/adjuvant therapy are allowed, but the time interval from the end of surgery to diagnosis of advanced or metastatic disease should be no less than 6 months;
5. Study sites must be able to provide relevant documentation of EGFR mutation and ALK fusion status of subjects which must be negative. If tumor tissue samples at or after the diagnosis of advanced tumors are available, archived within 1 year prior to the first dose or freshly obtained, testing for PD-L1 levels can be performed prior to enrollment or during the study;
6. Age ≥ 18 years;
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
8. Life expectancy of more than 3 months;
9. Adequate hematopoietic function, defined as absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109 /L, hemoglobin ≥ 90 g/L [no blood transfusion within 7 days or no erythropoietin (EPO) dependence];
10. Adequate liver function, defined as total bilirubin level ≤ 1.5 times the upper limit of normal (ULN); for patients without liver metastases, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN; for patients with documented liver metastases, AST and ALT levels ≤ 5 times ULN;
11. Adequate renal function, defined as serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); urine protein in urine routines less than 2+, if the patient has a urine protein ≥ 2+ at baseline, 24-hour urine should be collected and tested to ensure 24-hour urine protein quantification ≤ 1 g;
12. Adequate coagulation, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; anticoagulant therapy is allowed, as long as the PT is within the intended range of the anticoagulant drugs;
13. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of the study drug (Cycle 1, Day 1). If a urine pregnancy test cannot be confirmed as negative, a blood pregnancy test is required; women and men of childbearing potential must agree to use appropriate methods of contraception or have been surgically sterilized during the study and within 90 days after the last dose of the study drugs;
14. Able to comply with the study and follow-up procedures;
15. Sign the written informed consent prior to the implementation of any study-related procedures.

Exclusion Criteria Subjects who meet any of the following criteria are not eligible for inclusion in this study:

1. Mixed non-small cell and small cell carcinoma, or adenosquamous cell lung cancer with an adenocarcinoma component < 50% (if the adenocarcinoma component is ≥ 50%, the inclusion criteria are met);
2. Currently participating in an interventional clinical trial, or receiving other study drugs or treatment with study devices within 4 weeks prior to the first dose;
3. Patients who have received prior systemic anti-tumor therapy;
4. Patients who have received solid organ or blood system transplantation;
5. Active autoimmune disease requiring systemic therapy (e.g., use of disease modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Substitution therapy (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency, etc.) is not considered systemic therapy;
6. Diagnosis of immunodeficiency or ongoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study; physiologic doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent drugs) are allowed;
7. History of noninfectious pneumonitis requiring glucocorticoid therapy within 1 year prior to the first dose or current interstitial lung disease;
8. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive);
9. Untreated active hepatitis B; Note: subjects with hepatitis B who meet the following criteria are also eligible for inclusion:

   1. HBV viral load must be < 500 IU/ml prior to the first dose, and anti-HBV therapy should be administered at the discretion of the investigator throughout the study to avoid viral reactivation;
   2. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but viral reactivation needs to be closely monitored;
10. Subjects with active HCV infection (HCV antibody positive and HCV-RNA level higher than the lower limit of detection);
11. Pregnant and lactating women;
12. Known allergy to Camrelizumab, Pemetrexed, Carboplatin, or any of their excipients;
13. Malignancies other than NSCLC within 5 years prior to enrollment, except adequately treated cervical carcinoma in situ, basal cell or squamous epithelial cell skin carcinoma, localized prostatic carcinoma after radical surgery, and ductal carcinoma in situ after radical surgery.
14. Subjects with active pulmonary tuberculosis (TB) are excluded. Suspected active TB need to be excluded by chest x-ray, sputum examination and clinical symptoms and signs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial Objective Response Rate (iORR) | 1 year
  iORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response(PR: ≥30% decrease in the sum of diameters of target lesions) of intracranial lesion according to modified Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Intracranial Progression-Free Survival(iPFS) | 3.5year
  Intracranial Progression-free survival is defined as the duration from date of enrollment to the first occurrence of progression in intracranial lesions according to modified RECIST 1.1 or death from any cause
Objective Response Rate (ORR) | 3.5year
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Progression-free Survival (PFS) | 3.5year
  Progression-free survival is defined as the duration from date of enrollment to the first occurrence of progression of overall disease or death from any cause
Incidence of Adverse Events (AEs) | 3.5year
  Incidence of Adverse Events (AEs) in the treatment of Camrelizumab combined with pemetrexed / carboplatin for patients with brain metastasis according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Li-Kun Chen, MD., Principal Investigator — SunYat-sen University Cancer Center
Locations (1):
- Li-Kun Chen, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hou X, Zhou C, Wu G, Lin W, Xie Z, Zhang H, Yi J, Lv J, Cheng F, She F, Chen L. First-line camrelizumab plus pemetrexed and carboplatin for advanced non-squamous non-small-cell lung cancer with brain metastases (CAP-BRAIN): final results of a multicentre, open-label, single-arm, phase 2 trial in China. EClinicalMedicine. 2025 Nov 12;90:103638. doi: 10.1016/j.eclinm.2025.103638. eCollection 2025 Dec. PMID 41324015
- [Derived] Li M, Chen J, Yu H, Zhang B, Hou X, Jiang H, Xie D, Chen L. Cerebrospinal fluid immunological cytokines predict intracranial tumor response to immunotherapy in non-small cell lung cancer patients with brain metastases. Oncoimmunology. 2023 Dec 7;13(1):2290790. doi: 10.1080/2162402X.2023.2290790. eCollection 2024. PMID 38169917